CLINICAL TRIAL: NCT02947373
Title: PNOC 011: Pilot Study of Safety and Toxicity of Acquiring Hyperpolarized Carbon-13 Imaging in Children With Brain Tumors
Brief Title: Pilot Study of Safety and Toxicity of Acquiring Hyperpolarized Carbon-13 Imaging in Children With Brain Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Principal Investigator, Sabine Mueller, MD, PhD, Assistant Professor, University of California, San Francisco
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PNOC 011; 16088 (Other: University Of California, San Francisco HDCC)
Record Dates: First submitted 2016-10-24; First posted 2016-10-27 (Estimated); Last update posted 2021-06-24 (Actual); Status verified 2021-06

CONDITIONS: Pediatric Brain Tumors
Keywords: brain tumor; children
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Imaging Arm (Other): Patients will receive a one-time injection of Hyperpolarized Pyruvate prior to a single MR imaging examination that includes the acquisition of HP carbon-13 metabolic data.
  Interventions: Drug: Hyperpolarized Pyruvate

INTERVENTIONS:
Drug: Hyperpolarized Pyruvate — Hyperpolarized Pyruvate

SUMMARY:
This is a single arm pilot trial within the Pacific Pediatric Neuro-Oncology Consortium (PNOC).

The pilot study will look at the safety and toxicity of acquiring hyperpolarized carbon-13 imaging in children with brain tumors.

DETAILED DESCRIPTION:
This is an open label trial to assess the safety and tolerability of the adult tolerated dose of Hyperpolarized Pyruvate (HP) for metabolic imaging in children with brain tumors who do not require sedation for their MR imaging. Nine patients will receive a single MR imaging examination that includes the acquisition of hyperpolarized 13C metabolic data in combination with anatomic, diffusion, perfusion and lactate edited 1H spectroscopic imaging data. The data will be processed using custom designed software to estimate changes in levels of lactate/pyruvate and to relate them to abnormalities observed in the data from other MR modalities.

The results of this study will provide the safety data required to move this type of metabolic imaging into therapeutic trials to assess the utility of HP 13C lactate/pyruvate as a new surrogate marker of drug tumor penetration and early response to therapy in children with brain tumors.

ELIGIBILITY:
Inclusion Criteria:

* Children ≥ 3 years and ≤ 18 years of age with a diagnosis of a brain tumor and who do not require sedation for MR imaging
* Karnofsky ≥ 70 for patients ≥ 16 years of age, and Lansky ≥ 70 for patients < 16 years of age (See Appendix 1 Performance Status Criteria)
* Patients must not have any significant medical illnesses that in the investigator's opinion cannot be adequately controlled with appropriate therapy, would compromise the patient's ability to tolerate the imaging examination or any disease that will obscure toxicity or dangerously alter response to the imaging agent
* Patients must not be pregnant or breast feeding. Women of childbearing potential are required to obtain a negative pregnancy test within 14 days of starting treatment. Effective contraception (men and women) must be used in subjects of child-bearing potential
* Ability to understand and the willingness of the patient, parent or legal guardian to provide informed consent

Exclusion Criteria:

* Patients who are not able to comply with study and/or follow-up procedures
* Patients receiving active therapy on an investigational trial at the time of enrollment should consult with the study chair regarding potential interactions with other study agents. Patients who are enrolled in a clinical trial but are off- therapy and in follow up are eligible.
* Patients with history or evidence of cardiac dysfunction

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Actual)
Dates: Start 2017-01-25 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2020-07-31 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Adverse Events | 9 months
  Dose Limiting Toxicities will be assessed by monitoring for adverse events, scheduled laboratory assessments, vital sign measurements, ECGs, and physical examinations. The severity of the toxicities will be graded according to the NCI CTCAE v4.0. Adverse events and clinically significant laboratory abnormalities will be summarized by maximum intensity and relationship to study drug. Safety will be assessed during the infusion and at least for one hour after completion of the infusion as well as by phone 24 hours after the infusion. Descriptive statistics will be utilized to display the data on toxicity seen. Analyses will be performed for all patients having received at least one dose of study drug.

SECONDARY OUTCOMES:
Secondary analyses will include assessment of imaging quality, which will be descriptive in nature. | 12 months
  13C data will be acquired using the following sequence parameters;
  * a volumetric acquisition from a 4-5cm slice with 2D phase encoding and 1-D Echo-Planar Spectroscopic Imaging (EPSI) encoding, field of view (FOV) 20x24x10cm (1cc voxel size),
  * 1H scout; A further set of scout images will be obtained to re-establish appropriate landmarks.
  * High resolution anatomic imaging: These require a 3D localizing scan to define the graphical prescription;
  * Diffusion Images: This will be followed by diffusion tensor spin echo single shot echo planar images, 6 gradient directions, 22cm FOV, 128x128 matrix,
  * Lactate edited 3D magnetic resonance spectroscopic imaging (MRSI): water suppressed 1H magnetic resonance spectroscopy (MRS) with PRESS volume selection, out-of-voxel suppression with very spatially selective rf pulses, echo planar encoding in the signal intensity (SI) direction and 2D in-plane phase encoding

CONTACTS AND LOCATIONS:
Overall Officials: Sabine Mueller, MD, PhD, MAS, Study Chair — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No